CLINICAL TRIAL: NCT06877754
Title: Exploring the Effectiveness of Multimedia-Guided Self-Acupressure on Sanyinjiao (SP6) for Pain Relief in Young Women with Dysmenorrhea
Brief Title: Multimedia-Guided Self-Acupressure for Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, Taiwan (Other)
Responsible Party: Principal Investigator, Cheng, Jui-Fen, Associate Professor, China Medical University, Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMUH113-REC3-133
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Primary Dysmenorrhea, Acupressure, Sanyinjiao (SP6), Multimedia, Traditional Chinese Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimedia-Guided Acupressure at Sanyinjiao for Primary Dysmenorrhea (Experimental): Intervention: Self-Acupressure (Multimedia-Guided)
  Interventions: Behavioral: Self-Acupressure
- Control Group (No Intervention): The control group maintained their usual routines

INTERVENTIONS:
Behavioral: Self-Acupressure — Both groups received general health education videos. The experimental group performed SP6 acupressure starting one week before menstruation, 10 minutes per session, twice daily, until the fifth day of menstruation. The control group maintained their usual routines.
  Arms: Multimedia-Guided Acupressure at Sanyinjiao for Primary Dysmenorrhea

SUMMARY:
Background: Up to 84% of women of reproductive age experience primary dysmenorrhea, a gynecological issue. Approximately 15% of those affected by dysmenorrhea require sick leave from school or work due to severe pain, impacting both quality of life and causing substantial economic losses. Dysmenorrhea is typically categorized into primary and secondary types; this study focuses on primary dysmenorrhea. Primary dysmenorrhea occurs mainly during the ovulatory phase and is characterized by intense, crampy spasms, often accompanied by symptoms such as headaches, diarrhea, nausea, and vomiting. Acupressure massage is convenient, relatively safe, cost-effective, and can be enhanced through multimedia instruction to improve learning efficiency, accommodate individual needs, and overcome temporal and spatial limitations. Therefore, this study aims to investigate the effectiveness of multimedia-assisted acupressure at the Sanyinjiao acupoint for alleviating primary dysmenorrhea.

Purposes: To investigate the effectiveness of multimedia-guided acupressure at the Sanyinjiao acupoint in improving primary dysmenorrhea among young women.

Research method: This study employs a quasi-experimental pretest-posttest design over a three-month period. Participants will be recruited from two selected colleges in central Taiwan through voluntary enrollment. It is anticipated that each group, experimental and control, will consist of 22 participants. The experimental group will receive general multimedia health education videos along with self-made multimedia videos teaching acupressure at the Sanyinjiao acupoint. Treatment will commence one week before the menstrual cycle and continue until the 5th day of menstruation. On the other hand, the control group received general multimedia health education videos only.

Results: The data will be analyzed by SPSS 28.0 statistical software. Statistical methods will include descriptive statistics such as frequency, percentage, mean, and standard deviation analysis. Inferential statistics will include independent t-tests, chi-square tests, and paired t-tests to compare menstrual pain conditions before and after the intervention and the differences between the two groups.

DETAILED DESCRIPTION:
Background: Up to 84% of women of reproductive age experience primary dysmenorrhea, a gynecological issue. Approximately 15% of those affected by dysmenorrhea require sick leave from school or work due to severe pain, impacting both quality of life and causing substantial economic losses. Dysmenorrhea is typically categorized into primary and secondary types; this study focuses on primary dysmenorrhea. Primary dysmenorrhea occurs mainly during the ovulatory phase and is characterized by intense, crampy spasms, often accompanied by symptoms such as headaches, diarrhea, nausea, and vomiting. Acupressure massage is convenient, relatively safe, cost-effective, and can be enhanced through multimedia instruction to improve learning efficiency, accommodate individual needs, and overcome temporal and spatial limitations. Therefore, this study aims to investigate the effectiveness of multimedia-assisted acupressure at the Sanyinjiao acupoint for alleviating primary dysmenorrhea.

Purposes: To investigate the effectiveness of multimedia-guided acupressure at the Sanyinjiao acupoint in improving primary dysmenorrhea among young women.

Research method: This study employs a quasi-experimental pretest-posttest design over a three-month period. Participants will be recruited from two selected colleges in central Taiwan through voluntary enrollment. It is anticipated that each group, experimental and control, will consist of 22 participants. The experimental group will receive general multimedia health education videos along with self-made multimedia videos teaching acupressure at the Sanyinjiao acupoint. Treatment will commence one week before the menstrual cycle and continue until the 5th day of menstruation. On the other hand, the control group received general multimedia health education videos only.

Results: The data will be analyzed by SPSS 28.0 statistical software. Statistical methods will include descriptive statistics such as frequency, percentage, mean, and standard deviation analysis. Inferential statistics will include independent t-tests, chi-square tests, and paired t-tests to compare menstrual pain conditions before and after the intervention and the differences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1) Age: 18-30 years old; (2) Regular menstrual cycles (21-38 days); (3) Experienced dysmenorrhea in at least one of the past three months, with a self-reported pain score of >3 on the VAS scale.

Exclusion Criteria:

1. Diagnosed with pelvic organic diseases by a physician, such as endometriosis, adenomyosis, endometrial polyps, etc.;
2. Pregnant or breastfeeding women;
3. History of gynecological surgery;
4. Contraindications to acupoint massage, such as thrombocytopenia with bleeding tendency, local infection or inflammation at the massage site, excessive weakness, etc.;
5. Already capable of using acupoint massage to relieve pain;
6. Students enrolled in the course taught by the principal investigator.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-06 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) pain scores | 3 months
  using the VAS pain scores before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jui-Fen Cheng, Principal Investigator — China Medical University, China

IPD SHARING:
Plan to Share IPD: No